CLINICAL TRIAL: NCT03304613
Title: Resilience Skills Self-Management for Chronic Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Afton Hassett, Psy.D., Associate Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00124722; 5R01NR017096-05 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Spine Pain; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:2:1 as follows: e-CBT (n=120), PRISM (n=120) and usual care (n = 60).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Web-based Cognitive Behavioral Therapy (e-CBT) (Active Comparator): Patients randomized to e-CBT will undergo "Standard Web-based Cognitive Behavioral Therapy (e-CBT) Self-Management Program" and meet with a study medical assistant (MA) for an orientation session. The MA provides an overview of the program, explains the rationale for treatment, and directs them to the FibroGuide website. FibroGuide features the CBT modules that will be used by both groups. Patients will complete one module per week. Materials needed for the 8-week intervention including the instructions for each activity and forms for the written aspects of an activity (worksheets) will be provided in the first visit and available online. The FibroGuide website evolved from the evidence-based website Living Well with Fibromyalgia that has established efficacy for improving functional status and reducing pain.
  Interventions: Behavioral: Web-based Cognitive Behavioral Therapy (e-CBT) Self-Management
- Resilience-Enhanced web-based CBT Program (Experimental): Patients randomized to PRISM will undergo "Promoting Resilience through Innovative Self-Management" (PRISM) and meet with the MA for an orientation session. The MA describes the program, explains the rationale for treatment, and directs them to the FibroGuide and PRISM websites. Materials and worksheets are provided in the first visit and available online. The e-CBT elements retained are the core elements of CBT for pain, while the resilience-based activities capitalize on the best practices for positive activities interventions including having multiple overlapping activities, making favored activities standard practice beyond the study and having a coaching component.
  Interventions: Behavioral: Promoting Resilience through Innovative Self-Management
- Usual Care (No Intervention): Patients randomized to the usual care only group will have no contact with the study MAs. Usual care patients return for the same follow-up assessments (and electronic medical record review) at 8 weeks and at 6 and 12 months. Whereas major surgery including surgeries for pain, are exclusion criteria, spine and pain injections will be permitted.

INTERVENTIONS:
Behavioral: Web-based Cognitive Behavioral Therapy (e-CBT) Self-Management — Already noted.
  Arms: Standard Web-based Cognitive Behavioral Therapy (e-CBT)
Behavioral: Promoting Resilience through Innovative Self-Management — Already noted.
  Other Names: PRISM
  Arms: Resilience-Enhanced web-based CBT Program

SUMMARY:
The investigators will conduct a randomized controlled trial of an 8-week resilience-enhanced CBT online self-management program for chronic pain plus usual care (PRISM), standard e-CBT self-management plus usual care (e-CBT), and usual care alone. Thus, 300 individuals with chronic pain will undergo a comprehensive pre-intervention assessment that includes a blood draw (T1). Participants will then be randomized 2:2:1 as follows: e-CBT (n=120), PRISM (n=120) and usual care (n = 60). Immediately post-intervention (T2) and at 6 months (T3) and 12 months (T4) after that, participants undergo the same in-person assessment including blood draw. Telomerase activity will be assessed at T1, T2 and T3; and telomere length at T1 and T4

ELIGIBILITY:
Inclusion Criteria:

* Primary back or spine pain diagnosis from the Back & Pain Center at University of Michigan.
* High scores on the 2011 survey criteria for Fibromyalgia. The survey criteria for FM consist of an assessment of widespread pain and symptom severity.

Exclusion Criteria:

* Co-morbid autoimmune disorders, including rheumatoid arthritis and systemic lupus erythematosus.
* Medical conditions that can impair health status independent of spine pain and FM, including cardiopulmonary disorders (e.g. CHF, COPD), uncontrolled endocrine or allergic disorders (e.g., thyroid dysfunction, Type I diabetes), or malignancy within the preceding 2 years
* Current psychotic disorder (schizophrenia, etc.), dissociative identity disorder, untreated bipolar disorder, active suicide risk, or current alcohol / drug dependence.
* Planned major surgery in the next 12 months;
* Pregnancy or taking steroid medications
* Recent pain interventions ≤6 weeks prior to study (e.g., back surgery, epidural steroid injections) or planned interventions for the study period (e.g., surgery scheduled). Ongoing physical therapy will be allowed and new physical therapy or exercise regimen will be addressed during data analysis;
* Cognitive impairment or dementia (inability to give consent or meaningfully participate);
* Pending or recently received (within 1 years) pain-related disability or Workman's Compensation;
* Unable to read or fluently converse in English;
* Planning to move from the area in next 14 months;
* In the judgment of the PIs the individual would not be able to meaningfully participant.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire-Revised (FIQ-R) | At 8-week assessment point
  The Fibromyalgia Impact Questionnaire-Revised (FIQR) assesses the total spectrum of problems and responses to therapy. The 2009 revised version contains 21 items assessing broad domains such as physical function, overall impact, and a wide range of symptoms. The measure is self-report with a recall period of the past week and requires only several minutes to complete.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | At 8-week assessment point
  The BPI is a 15-item self-report measure that has been validated for use in a wide variety of pain states. The BPI assesses for the presence of pain, pain intensity (i.e., worst, least, average, current) and functional interference from pain.
Pittsburgh Sleep Quality Index (PSQI) | At 8-week assessment point
  The PSQI is a widely used, valid and reliable measure of global sleep quality and sleep-related symptoms.149 The 19-items yield 7 component-scores that reflect common sleep problems such as subjective sleep quality, sleep disturbance and use of sleep medication.
PROMIS Fatigue-Short Form | At 8-week assessment point
  The PROMIS Fatigue-Short Form consists of 8 items that assess the impact and experience of fatigue in the past week. It uses a 5-point Likert-like scale with response options that range from "Not at all" to "Very much." A raw score is calculated by summing scores across items then a conversion table is used to calculate T-scores with higher scores indicating greater fatigue.
Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | At 8-week assessment point
  The MISCI is a 10-item measure based upon items developed for PROMIS that assesses perceived difficulties within 5 domains: mental clarity, memory, language, executive functioning, and attention/concentration.
Subjective well-being | At 8-week assessment point
  Subjective well-being has at least three components: positive affective appraisal, negative affective appraisal, and life satisfaction. Composite scores for well-being will be calculated using scores obtained on Positive and Negative Affect Schedule (PANAS) and the Satisfaction with Life Scale (SWLS).
Pain Catastrophizing Scale (PCS) | At 8-week assessment point
  . Catastrophizing will be measured using the Pain Catastrophizing Scale (PCS).144 The PCS contains 13 statements regarding various beliefs about pain. A total score is obtained by summing the responses to all items.
Patient Health Questionnaire 9-item (PHQ-9): | At 8-week assessment point
  The PHQ-9 is a 9-item multipurpose instrument that has utility for screening, diagnosing, monitoring, and measuring the severity of depression.
Generalized Anxiety Disorder 7-item (GAD-7) | At 8-week assessment point
  The GAD-7 is a 7-item measure of anxiety. It has good reliability, criterion, construct, and factorial validity. It has a sensitivity of 89% and specificity of 82% for generalized anxiety disorder.
Perceived Stress Scale (PSS) | At 8-week assessment point
  The 10-item PSS will be used evaluate an individual's assessment of stress. Participants rate stress on a numeric rating scale from 0 to 10 where higher scores reflect higher levels of stress. Total scores range from 0 to 100.
Six-Minute Walk Test (6MWT) | At 8-week assessment point
  The 6MWT measures the distance a participant is able to walk over a total of six minutes on a hard, flat surface. Participants are instructed to walk as far as possible, but allowed to self-pace and rest as needed.
Sit-to-Stand Test | At 8-week assessment point
  Patients are instructed to stand up 5 times from a chair without arms as fast as possible. The test is repeated twice as this improves reliability. Average time is calculated in seconds.
Telomerase activity as measured by the Droplet Digital PCR (ddPCR) method | At 8-week assessment point
  The Blackburn lab collaborated with Biorad to develop a highly sensitive, quantitative and high throughput droplet digital PCR (ddPCR) method to measure telomerase activity in unstimulated PBMCs. This new method has over 10-fold increased sensitivity and over 5-fold increased throughput compared to the currently used gel method.
Telomere length | At 1 year assessment point
  The DNA will then be analyzed for telomere length using a quantitative polymerase chain reaction (PCR) measurement assay adapted from the methods described by Cawthon with modifications by Lin (Co-I).

CONTACTS AND LOCATIONS:
Locations (1):
- Back & Pain Center, University of Michigan, Ann Arbor, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT03304613/ICF_000.pdf